CLINICAL TRIAL: NCT06868459
Title: Pressure-enabled Retrograde Occlusive Therapy With Embolization for Control of Thyroid Disease (PROTECT Registry): A Multicenter Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Sarasota Memorial Health Care System (Other)
Collaborators: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Juan C. Camacho, MD, Principal Investigator, Sarasota Memorial Health Care System
Other Study IDs: 24-ENT-97
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Hyperthyroidism; Goiter; Multinodular Goiter; Thyroid Nodules; Thyroid Disease; Hyperthyroidism; Toxic Multinodular Goiter
Keywords: PED-TAE; TriNav Infusion System; Thyroid artery embolization
MeSH Terms: conditions — Hyperthyroidism; Goiter; Thyroid Nodule; Thyroid Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who have undergone PED-TAE using the TriNav Infusion System at participating study sites.: Subjects with planned PED-TAE delivered via TriNav will receive their treatment following routine standard of care procedures. Post-procedural data obtained by a patient chart review will be collected in a study database. No additional study-specific interventions or visits outside of the routine clinical treatment will be performed.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Subjects with planned PED-TAE delivered via TriNav will receive their treatment following routine standard of care procedures. Post-procedural data obtained by a patient chart review will be collected in a study database. No additional study-specific interventions or visits outside of the routine clinical treatment will be performed.

SUMMARY:
Multi-center registry study to evaluate disease-related quality of life outcomes of thyroid embolization via pressure-enabled delivery (PED-TAE). Additional technical success data on parenchymal volume reduction, thyroid function tests changes and post-procedural complications will be recorded. Data will be collected for patients who have undergone PED-TAE using the TriNav Infusion System at participating sites. The registry study will include up to 10 sites, with Sarasota Memorial Health Care System acting as the lead site responsible for maintaining and monitoring the study database.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years and or older and 89 years or younger
2. Having undergone PED-TAE using the TriNav Infusion System
3. Meeting one of the following criteria:

   1. Documented subclinical and or clinical hyperthyroidism in the presence of a toxic multinodular goiter or a toxic nodule > 20 ml
   2. Patients' ineligible or refusing surgery, radio-iodine therapy or percutaneous ablation
   3. Non-functioning multinodular goiters or nodule causing compressive symptoms including but not limited to neck pain, dysphagia, stridor, exercise induced dyspnea and/or pressure symptoms
   4. Bethesda category 2-3 (benign, or atypia or follicular lesion of undetermined significance) on 2 separate fine-needle aspiration biopsy (FNAB) results with a benign molecular profile with patient declining surgical resection

Exclusion Criteria:

1. Renal insufficiency
2. Unable to tolerate angiography including pregnancy and severe allergy to contrast media
3. Bethesda 4-6 on FNAB (suspicious for follicular neoplasm, suspicious for malignancy, or malignant)
4. <18 years old or >89 years old
5. Graves' disease or inflammatory thyroiditis (Hashimoto's) or other condition with the presence of an extensive collateral network as demonstrated or initial angiography
6. Presence of a bovine arch or any other anatomical variant with no inferior thyroid artery present
7. Prior thyroid thermal ablation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that may be included in the registry study are those who have undergone PED-TAE using TriNav at the selected study sites. Data will be collected on patients meeting eligibility criteria.
  Study subjects will not be informed of their inclusion in this registry dataset, and the results of this research will not be reported to study subjects at the conclusion of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
ThyPro-39 questionnaire | 6 months
  Change in quality of life as measured by ThyPro-39 questionnaire at 6-months (+/- 60). Responses to each statement are measured on a Likert scale ranging from '0= no symptoms or problems' to '4= severe symptoms or problems' based on the period of the last 4 weeks. Higher scores indicate greater impact on quality of life due to thyroid issues.
Procedure related adverse events | 6 months
  Safety as measured by the rate of procedure related adverse events as measured by SIR criteria at 2-weeks (+/- 7 days), 3- (+/- 30 days) and 6-months (+/- 60 days) post PED-TAE using TriNav treatment.

SECONDARY OUTCOMES:
Thyroid volume change | 6 months
  Thyroid volume change based on 3D CT volumetry at 6-months (+/- 60 days) post-treatment
Change in TSH, T3 and T4 | 6 months
  Change in TSH, T3 and T4 levels at 2-weeks (+/- 7 days), 3-(+/- 30 days) and 6-months (+/- 60 days) post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tamela Fonseca, PhD, RN, CCRC, NE-BC, Study Director — Sarasota Memorial Health Care System
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yilmaz S, Habibi HA, Yildiz A, Altunbas H. Thyroid Embolization for Nonsurgical Treatment of Nodular Goiter: A Single-Center Experience in 56 Consecutive Patients. J Vasc Interv Radiol. 2021 Oct;32(10):1449-1456. doi: 10.1016/j.jvir.2021.06.025. Epub 2021 Jul 10. PMID 34256121
- [Background] Wiener JD, de Vries AA. On the natural history of Plummer's disease. Clin Nucl Med. 1979 May;4(5):181-90. doi: 10.1097/00003072-197905000-00002. PMID 582300
- [Background] Watt T, Cramon P, Hegedus L, Bjorner JB, Bonnema SJ, Rasmussen AK, Feldt-Rasmussen U, Groenvold M. The thyroid-related quality of life measure ThyPRO has good responsiveness and ability to detect relevant treatment effects. J Clin Endocrinol Metab. 2014 Oct;99(10):3708-17. doi: 10.1210/jc.2014-1322. Epub 2014 Jul 8. PMID 25004246
- [Background] Sjolin G, Watt T, Bystrom K, Calissendorff J, Cramon PK, Nystrom HF, Hallengren B, Holmberg M, Khamisi S, Lantz M, Planck T, Torring O, Wallin G. Long term outcome after toxic nodular goitre. Thyroid Res. 2022 Nov 1;15(1):20. doi: 10.1186/s13044-022-00138-0. PMID 36316779
- [Background] Russell JO, Desai DD, Noel JE, Hussein M, Toraih E, Seo S, Wolfe S, Omar M, Issa P, Orloff LA, Tufano RP, Kandil E. Radiofrequency ablation of benign thyroid nodules: A prospective, multi-institutional North American experience. Surgery. 2024 Jan;175(1):139-145. doi: 10.1016/j.surg.2023.07.046. Epub 2023 Nov 10. PMID 37953141
- [Background] Roque C, Santos FS, Pilli T, Dalmazio G, Castagna MG, Pacini F. Long-term Effects of Radioiodine in Toxic Multinodular Goiter: Thyroid Volume, Function, and Autoimmunity. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa214. doi: 10.1210/clinem/dgaa214. PMID 32320467
- [Background] Paschke R. Molecular pathogenesis of nodular goiter. Langenbecks Arch Surg. 2011 Dec;396(8):1127-36. doi: 10.1007/s00423-011-0788-5. Epub 2011 Apr 14. PMID 21487943
- [Background] Moon JH, Hyun MK, Lee JY, Shim JI, Kim TH, Choi HS, Ahn HY, Kim KW, Park DJ, Park YJ, Yi KH. Prevalence of thyroid nodules and their associated clinical parameters: a large-scale, multicenter-based health checkup study. Korean J Intern Med. 2018 Jul;33(4):753-762. doi: 10.3904/kjim.2015.273. Epub 2017 Jul 7. PMID 28859466
- [Background] Elte JW, Bussemaker JK, Haak A. The natural history of euthyroid multinodular goitre. Postgrad Med J. 1990 Mar;66(773):186-90. doi: 10.1136/pgmj.66.773.186. PMID 2114018
- [Background] Dean DS, Gharib H. Epidemiology of thyroid nodules. Best Pract Res Clin Endocrinol Metab. 2008 Dec;22(6):901-11. doi: 10.1016/j.beem.2008.09.019. PMID 19041821
- [Background] Cheng KL, Liang KW, Lee HL, Wang HY, Shen CY. Thyroid artery embolization of large solitary symptomatic benign thyroid nodules through transradial approach. Quant Imaging Med Surg. 2023 Aug 1;13(8):5355-5361. doi: 10.21037/qims-22-1385. Epub 2023 May 30. PMID 37581037
- [Background] Campenni A, Avram AM, Verburg FA, Iakovou I, Hanscheid H, de Keizer B, Petranovic Ovcaricek P, Giovanella L. The EANM guideline on radioiodine therapy of benign thyroid disease. Eur J Nucl Med Mol Imaging. 2023 Sep;50(11):3324-3348. doi: 10.1007/s00259-023-06274-5. Epub 2023 Jul 3. PMID 37395802
- [Background] Berghout A, Wiersinga WM, Smits NJ, Touber JL. Interrelationships between age, thyroid volume, thyroid nodularity, and thyroid function in patients with sporadic nontoxic goiter. Am J Med. 1990 Nov;89(5):602-8. doi: 10.1016/0002-9343(90)90178-g. PMID 2239979
- [Background] Bahre M, Hilgers R, Lindemann C, Emrich D. Thyroid autonomy: sensitive detection in vivo and estimation of its functional relevance using quantified high-resolution scintigraphy. Acta Endocrinol (Copenh). 1988 Feb;117(2):145-53. doi: 10.1530/acta.0.1170145. PMID 2837884